CLINICAL TRIAL: NCT04903340
Title: Assessment of the Impact of Acquisition Time, Respiratory Gating and New Qclear Reconstruction Modalities on the Quantification of Dosimetry in Selective Internal Radiotherapy
Acronym: PYR
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/60
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PET/CT Exam — PET/CT image processing application of reconstruction parameters: scan time, respiratory gating, Q-clear

SUMMARY:
Post-processing of Positron Emission Tomography (PET) acquired images, performed following radioembolization treatment with microspheres at 90Y in hepatocellular carcinoma patients, is subject to changes commercialized by General Electric : respiratory motion correction, specific reconstruction algorithms. We propose to test the possible combinations of these reconstruction parameters to determine which ones to apply for an optimal quality exam with the shortest scan time possible

ELIGIBILITY:
Inclusion Criteria:

* patient with hepatocellular carcinoma
* with radioembolization treatment decided
* over the age of 18

Exclusion Criteria:

* radiembolization not possible
* acquisition of PET/CT imaging at 90Y not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Average dose value (Gy) of tumor liver and healthy liver obtained according to reconstruction configuration. | Day 0 (PET/CT Exam)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided